CLINICAL TRIAL: NCT02533349
Title: Randomized Controlled Trial of Proton Pump Inhibitor With Prokinetics or Placebo in Patients With Laryngopharyngeal Reflux Disease
Brief Title: Trial of Proton Pump Inhibitor With Prokinetics or Placebo in Patients With Laryngopharyngeal Reflux Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Man Ki Chung, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-05-007-001
Record Dates: First submitted 2015-08-04; First posted 2015-08-26 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Laryngopharyngeal Reflux Disease
Keywords: laryngopharyngeal reflux disease; prokinetics; proton pump inhibitor
MeSH Terms: interventions — Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proton pump inhibitor + prokinetics (Active Comparator): Patient will be prescribed proton pump inhibitor (pantoprazole, 40mg, 1T QD) with prokinetics (Motilitone, 30mg, 1T, TID) for 3months.
  Interventions: Drug: Motilitone; Drug: Pantoprazole
- Proton pump inhibitor + placebo (Placebo Comparator): Patient will be prescribed proton pump inhibitor (pantoprazole, 40mg, 1T QD) with placebo (Motilitone, 30mg, 1T, TID) for 3months.
  Interventions: Drug: Pantoprazole; Drug: Placebo

INTERVENTIONS:
Drug: Motilitone — 30mg, 1 tablet, 3 times a day
  Arms: Proton pump inhibitor + prokinetics
Drug: Pantoprazole — 40mg, 1 tablet, 1time a day
Drug: Placebo — 30mg, 1 tablet, 3 times a day
  Arms: Proton pump inhibitor + placebo

SUMMARY:
Based on meta-analysis of prokinetics trials in laryngopharyngeal reflux disease (LPRD) (Glicksman et al. 2014), well designed study was performed in 4 articles. But, those studies had several problems including inclusion criteria, randomization methods, and placebo medication. They had similar results that prokinetics and proton pump inhibitor (PPI) had synergistic effect for management of LPRD. Therefore, the aim of study is to evaluate the efficacy of prokinetics as an additional medication to proton pump inhibitor by well designed randomized double blind case-control study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65 years
* Reflux Symptom Index (RSI) > 7 and, Reflux Finding Score (RFS) > 13

Exclusion Criteria

* Taken proton pump inhibitor within 3months
* Taken steroid within 3months
* Pregnancy
* Breast feeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Reflux symptom index (questionnaire) | 1 month after medication
  Reflux symptom index is validated questionnaire for laryngopharyngeal reflux disease. It consists of 9 items, and scale of each item ranges from 0 to 5 with maximal total score of 45.
Reflux finding score (scoring of laryngeal stroboscopy finding score) | 1 month after medication
  Reflux finding score is an 8-item clinical severity scale based on findings during laryngeal stroboscopy. The scale ranges from 0 (no abnormal findings) to a maximum of 26 (worst score possible).

SECONDARY OUTCOMES:
Reflux symptom index (questionnaire) | 3 months after medication
  Reflux symptom index is validated questionnaire for laryngopharyngeal reflux disease. It consists of 9 items, and scale of each item ranges from 0 to 5 with maximal total score of 45.
Reflux finding score (scoring of laryngeal stroboscopy finding score) | 3 months after medication
  Reflux finding score is an 8-item clinical severity scale based on findings during laryngeal stroboscopy. The scale ranges from 0 (no abnormal findings) to a maximum of 26 (worst score possible).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Result] Glicksman JT, Mick PT, Fung K, Carroll TL. Prokinetic agents and laryngopharyngeal reflux disease: Prokinetic agents and laryngopharyngeal reflux disease: a systematic review. Laryngoscope. 2014 Oct;124(10):2375-9. doi: 10.1002/lary.24738. Epub 2014 Jun 10. PMID 24782414